CLINICAL TRIAL: NCT05737264
Title: Safety and Effectiveness of Transcatheter Treatment of Severe Native Aortic Regurgitation With Self-Expandable Valve Implantation: a Multicenter, Observational,Cohort Study(SENSE-AR)
Brief Title: TAVR in Adults With Pure Severe Aortic Regurgitation
Acronym: SENSE-AR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-518-01
Record Dates: First submitted 2023-01-29; First posted 2023-02-21 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-01

CONDITIONS: Transcatheter Aortic Valve Replacement; Aortic Regurgitation
Keywords: Transcatheter Aortic Valve Replacement; Aortic Regurgitation; Observational
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVR group: The group that undergoes transcatheter aortic valve replacement

SUMMARY:
The study aimed to evaluate the efficacy and safety of transcatheter aortic valve replacement (TAVR) in patients with severe native valve aortic insufficiency. It is a multicentre, observational cohort study. The primary endpoint consisted of a composite of all-cause death, disabling stroke, or rehospitalization for heart failure at 12 months postoperatively. According to previous research results and opinions of expert groups, the sample size was expected to be 76 cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Patients with severe aortic regurgitation (> grade 3) diagnosed by transthoracic echocardiography should meet any of the following conditions for semi-quantitative assessment of the degree of aortic regurgitation and any condition for quantitative assessment of the degree of aortic regurgitation: (1) semi-quantitative assessment of the degree of aortic regurgitation: aortic regurgitation bundle width/left ventricular outflow tract diameter ≥ 65%; or aortic regurgitation neck width > 6 mm; or full-diastolic blood flow reflux in the proximal abdominal aorta; (2) quantitative assessment of the degree of aortic regurgitation: aortic regurgitation volume ≥ 60 ml/beat; or aortic regurgitation fraction ≥ 50%; or effective regurgitation orifice area ≥ 0.3 cm2
* TAVR has been performed;
* Patients can understand and voluntarily participate in this clinical study, sign informed consent, and adhere to clinical follow-up.

Exclusion Criteria:

* History of aortic valve replacement;
* Combined with moderate-severe mitral regurgitation and moderate aortic stenosis;
* Acute endocarditis or other acute cardiac inflammation;
* Allergic or contraindicated to related drugs (aspirin, clopidogrel, warfarin, contrast agent);
* Other conditions judged by the investigator as not suitable for the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic regurgitation undergo transcatheter aortic valve replacement in medical centers
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 12 months
  Death caused by any reason
Disabling stroke | 12 months
  Stroke that results in a disabled state
Rehospitalization for heart failure | 12 months
  Rehospitalization for heart failure

SECONDARY OUTCOMES:
Device success | intraoperative
  Absence of procedural mortality AND Correct positioning of a single prosthetic heart valve into the proper anatomical location AND Intended performance of the prosthetic heart valve (no prosthesis- patient mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s, AND no moderate or severe prosthetic valve regurgitation)
Perioperative complications | up to 1 week
  Perioperative complications conclude Life-threatening bleeding, Acute kidney injury-Stage 2 or 3 (including renal replacement therapy), Coronary artery obstruction requiring intervention, Major vascular complications, and Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
New permanent pacemaker implantation(PPI) | up to 1 week
  New PPI indications:
  1. persistent high-degree AV block
  2. sick sinus syndrome
New complete left bundle branch block(CLBBB) | up to 1 week
  Diagnostic criteria are defined as follows:
  1. Rhythm must be of super-ventricular origin (EG: ventricular activation coming from atrial or AV nodal activation)
  2. QRS Duration greater than 120 ms
  3. Lead V1 should have either a QS or a small r wave with large S wave
  4. Lead V6 should have a notched R wave and no Q wave.
Valve-related dysfunction | 12 months
  Mean aortic valve gradient ≥20 mmHg, EOA ≤0.9-1.1 cm and DVI <0.35 m/s, and/or moderate or severe prosthetic valve regurgitation, and/or Prosthetic valve endocarditis, and/or Prosthetic valve thrombosis
NYHA class Ill or IV | 12 months
  The New York Heart Association (NYHA) class Ill or IV

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China